CLINICAL TRIAL: NCT04684069
Title: "Syringe Free" Long-Axis In-Plane vs. Short-Axis Out-of-Plane Approach for Ultrasound-Guided Central Venous Catheter Placement in Critically Ill Children: A Prospective Randomized Study
Brief Title: "Syringe Free" Long-Axis In-Plane vs. Short-Axis Out-of-Plane Approach for Central Venous Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AtaturkCatheter
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Catheter Complications; Critical Illness
Keywords: ultrasound; catheter; long axis; short axis; pediatrics; syringe free
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- syringe free long axis in-plane (Active Comparator)
  Interventions: Device: Long-axis syringe free in-plane
- Short axis out-of-plane (Sham Comparator)
  Interventions: Device: Short-axis out-of-plane

INTERVENTIONS:
Device: Long-axis syringe free in-plane — Long-axis syringe-free in-plane catheter placement
  Arms: syringe free long axis in-plane
Device: Short-axis out-of-plane — Short-axis out-of-plane catheter placement
  Arms: Short axis out-of-plane

SUMMARY:
Internal jugular, subclavian, or femoral veins are often used for central venous catheter (CVC) placement. Regardless of which vein is preferred, the "Seldinger" technique is used most frequently. The most commonly used method with ultrasound is the short-axis out-of-plane approach. The main problem in this method is that the correct needle tip is missed, and it causes some complications by causing posterior wall punctures. The "Syringe-free" technique is first reported by Matias et al. in adults; it is a technique that allows full real-time monitoring of the guidewire insertion into the vein without blood aspiration. It is a great advantage in CVC placement, especially with the long-axis in-plane approach. When the literature is reviewed, no study other than a 12 case study in which brachiocephalic vein catheterization related to CVC placement was performed using this technique in children was found. There is no randomized study comparing the "Syringe-free" Long-Axis In-Plane technique with the classic Short-Axis Out-of-Plane technique in pediatric patients.

This study compares these two techniques' efficacy and complication rates in critically ill children requiring CVC placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 3 months, younger than 15 years old
* Critical illness pediatrics

Exclusion Criteria:

* Patients younger than 3 months and older than 15 years,
* body weight less than 5000 gr,
* anatomical malformation in the neck,
* infection at the intervention site,
* thrombosis

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Performing time | First 10 minutes
  The time between the insertion of the needle through the skin and insertion of the guidewire into the internal jugular vein.

SECONDARY OUTCOMES:
Complications | First 24 hours
  Catheter related complications
Number of neddle pass | First 10 minutes
  a change in needle direction without pulling the entire needle out of the skin
First pass success | First 10 minutes
  Successful catheterization with only one needle pass.
New puncture | First 10 minutes
  Withdraw the needle from the skin to change the puncture site

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaban O, Turgut M, Aydin T. Ultrasound-guided supraclavicular brachiocephalic vein catheterization in children: Syringe-free in-plane technique with micro-convex probe. J Vasc Access. 2020 Mar;21(2):241-245. doi: 10.1177/1129729819867221. Epub 2019 Sep 6. PMID 32174238
- [Background] Matias F, Semedo E, Carreira C, Pereira P. [Ultrasound-guided central venous catheterization - "Syringe-Free" approach]. Rev Bras Anestesiol. 2017 May-Jun;67(3):314-317. doi: 10.1016/j.bjan.2016.08.005. Epub 2016 Sep 17. Portuguese. PMID 27650385